CLINICAL TRIAL: NCT07170566
Title: The Use of a Decellularised Porcine Placental Extracellular Matrix in Hard-to-heal Wounds: A Retrospective, Observational Study of the Real-world Safety and Performance of InnovaMatrix® AC at a Single Centre
Brief Title: A Retrospective, Observational Study of the Real-world Safety and Performance of InnovaMatrix® AC at a Single Centre
Status: Completed | Type: Observational
Sponsor: ConvaTec Inc. (Industry)
Collaborators: Charleston Wound Care Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: WC-23-444
Record Dates: First submitted 2025-08-21; First posted 2025-09-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Wound Heal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with Hard to Heal Wounds Who are Treated with InnovaMatric AC: Adult subjects seen at the study site between 1 May 2022 (the date of first product use according to the study site) to 27 March 2024 (the date of contract signature), who meet the inclusion and exclusion criteria. There will be no new patient visits associated with this retrospective study, therefore patient duration is not applicable.
  Interventions: Device: innovaMatrix AC

INTERVENTIONS:
Device: innovaMatrix AC — nnovaMatrix® AC consists of ECM derived from porcine placental material. The device is supplied in a variety of sterile sheet configurations. It is packaged in double peel-open packages and is intended for single use only. The device is terminally sterilised using E-Beam sterilisation and is for licensed healthcare practitioner use only.
  InnovaMatrix® AC is composed of collagen, elastin, laminin, fibronectin, hyaluronic acid and sulphated glycosaminoglycans. The wound dressing is provided in sheets that are approximately 40-100 microns thick in sizes ranging from 1 x 1cm to 5 x 5cm. They are provided as single-use, sterile wound coverings.
  InnovaMatrix® AC received Food and Drug Administration (FDA) clearance under K193552 on October 21, 2020. InnovaMatrix® AC has an FDA classification of KGN, which designates it as a collagen wound dressing.

SUMMARY:
The use of a decellularised porcine placental extracellular matrix in hard-to-heal wounds: A retrospective study of the real-world performance of InnovaMatrix® AC at a single centre.

DETAILED DESCRIPTION:
Hard-to-heal wounds are defined as wounds that do not transition through the normal phases of healing in a timely manner.1 With a global prevalence of ~1.9 per 1000, it is predicted that the incidence will increase with the ageing population.2-5 Furthermore, hard-to-heal wounds are associated with a significant reduction in health-related quality of life and place a great burden on healthcare systems.4,6-9 In the UK, the annual National Health Service cost of wound management in 2017/2018 was £8.3 billion; £2.7 billion and £5.6 billion were associated with managing healed and unhealed wounds, respectively.5 Moreover, wound care accounts for 2-4% of healthcare expenditure in Europe and costs $28 billion USD per year in the US.7-11

Specifically, the cost of care for diabetic patients with a diabetic foot ulcer (DFU) vs. those without a DFU is 5.4 times higher in the year after first diagnosis while costs for treatment of highest grade ulcers are 8 times higher than low-grade ulcers.12 Use of advanced therapies, while sometimes costly, have been shown to reduce long-term costs, including reduced foot complications and lower amputation rates.12 In 1998, Holzer et al conducted a retrospective analysis of the costs for lower extremity ulcers in patients with diabetes and concluded that, given the high costs associated with treating these ulcers, the development of better treatment strategies is warranted.13 One such advanced therapy in the treatment of chronic wounds is the use of Cellular, Acellular and Matrix-like products (CAMPs). These materials have been used successfully for many years in the treatment of hard-to-heal wounds, as well as other applications including soft tissue repair, tendon/ligament repair, plastic/reconstructive surgeries, and urological surgery.

In wound care, CAMPs were developed as an alternative to skin grafts in the management of hard-to-heal wounds. They are derived from either natural or synthetic sources, which provide an artificial extracellular matrix (ECM) that allows for infiltration of host cells. Natural sources include human cadaver skin processed to remove the cellular components and retain the structural proteins of the dermis, and collagen obtained from bovine and porcine sources. Synthetic sources include various degradable polymers.

Numerous studies have explored the safety and performance of CAMPs. Kavros, et.al. performed a prospective, multicentre study that included 71 patients to evaluate the usage of PriMatrix® for diabetic foot ulcers.14 Sixteen patients failed to meet inclusion and exclusion criteria so only 55 patients were enrolled in the intent-to-treat (ITT) population. A total of 46 patients completed the 12-week study period. Thirty-five of the 46 patients (76%) were healed at 12 weeks and the patients that were not completely healed had a reduction in wound area of 71.4% at 12 weeks. One of the ITT patients discontinued from the study had a complication related to the wound in the study. The authors concluded," the results from this multicentre perspective study demonstrate that PriMatrix® coupled with debridement, moist wound therapy, and pressure offloading is a successful strategy to heal chronic DFUs."14

Frykberg, et.al. executed a multi-centre randomised clinical trial to compare the efficacy of MatriStem MicroMatrix and MatriStem Wound Matrix to Dermagraft in the management of non-healing diabetic foot ulcers.15 Fifty-six patients were randomised in a 1:1 ratio between the two treatment groups. No statistical difference in demographic make-up was observed between the treatment groups. Wound measurements were assessed using a digital wound measurement system. All subjects completed a Patient-Reported Outcome Measures (PROMs) questionnaire at multiple time points during the study. The results of the interim analysis did not demonstrate a statistical difference in wound outcomes between the two study products but there was a significant difference in treatment costs favouring MatriStem.15

Dorman, et.al. performed a retrospective review of four patients treated with MatriStem for the treatment of wounds associated with pilonidal disease.16 The treatments varied slightly by patient but generally involved the use of MatriStem MicroMatrix for the deep areas of the wound and then a sheet version. The sheet versions included multilayer, fenestrated, six layer and dual layer configurations. All four patients achieved full closure of the wounds at a mean of 51 days.16

Rommer, et.al. detailed their experience with MatriStem for large non-healing wounds from radiation burns.17 The three patients presented were each treated with a combination of MatriStem MicroMatrix and MatriStem Wound Matrix. The initial wound for the first patient was 5cm x 7cm, the initial wound for the third patient was 6cm x 6cm, and the initial wound for the second patient was not reported. All three patients had successful wound closure between 6 and 16 weeks with continued closure from multiple years.17

The Lullove retrospective review of twenty-nine patients with 34 wounds examined the treatment of chronic non-healing wounds with meshed PriMatrix.18 The types of wounds treated included diabetic ulcers, venous stasis ulcers, nonhealing traumatic wounds, other non-healing wounds, including tunnelling and undermined wounds. The wounds treated in the study had an average area of 19.6 square centimetres and a maximum area of 39.1 square centimetres. Wounds of different types and sizes healed in 10 to 15 weeks with 1.2 to 2.6 applications of PriMatrix.18

One such CAMP and the focus of this study is InnovaMatrix® AC, a decellularised ECM topical wound covering derived from porcine placental tissue harvested, according to Good Manufacturing Practices, by Tissue Source, LLC, in Lafayette, Indiana. Convatec Triad Life Sciences, in Memphis, Tennessee, processes the tissue into the ECM topical wound coverings. The composition of InnovaMatrix® AC includes the amnion and chorion from the porcine placenta.

The safety and performance of the predicate device for InnovaMatrix® AC, Oasis® Wound Matrix, has been investigated by multiple studies.

Brown-Etris, et.al. performed a randomised multicentre clinical trial of 130 patients with chronic pressure ulcers treated with Oasis® Wound Matrix and standard care versus standard care only.19 The percentage of patients completely healed in the Oasis group versus control was trending towards significance (p=0.111) but the percentage of Oasis versus control patients with 90% reduction in ulcer surface area was significantly higher (p=0.037). There was no difference in complication reported between the two groups. The study concluded that the addition of Oasis® Wound Matrix to standard care increases the incidence of 90% reduction in ulcer surface area.19

Romanelli, et.al. treated 50 patients with arterial/venous or venous only ulcers of the lower leg.20 The patients were randomised to either Oasis® Wound Matrix or standard moist wound dressing. The Oasis treated group healed, on average, at 5.4 weeks compared to 8.3 weeks for the standard moist dressing group {p=0.02). No adverse events were noted in either group. The authors concluded that Oasis had significantly better healing rates within 8 weeks as compared with conventional moist wound dressing.20

Baldursson, et.al. conducted a parallel-group, double-blinded, randomised controlled trial to compare Kerecis Omega3 Wound to Oasis® Wound Matrix for the treatment of wounds.21 Healthy volunteers had two 4mm full thickness punch wounds made 2cm apart on their non-dominant arm. The wounds were assessed by a dermatologist on days 1, 7, 14, 21 and 28. The wounds were treated with either Kerecis Omega3 Wound or Oasis® Wound Matrix according to the randomisation design. The primary endpoint was healing at 28 days which was defined as full epithelialisation. At 28 days, 76 of 80 wounds (95%) in Kerecis treated patients and 79 of 82 wounds (96.3%) in Oasis treated patients had healed. Statistical analysis demonstrated that Kerecis was non-inferior to Oasis in wound healing. Adverse events, including mild erythema and irritation, were noted in a small number of patients and within the limits expected and described in similar studies.21

Niezgoda, et.al. conducted a prospective, randomised, controlled multi-centre clinical trial that compared Oasis® Wound Matrix with Regranex Gel in the treatment of diabetic foot ulcers.22 Thirty-seven patients were randomised to Oasis treatment while thirty-six received Regranex gel. A secondary dressing was also applied to all patients following placement of the test article. The wounds were cleaned and debrided, as needed, during weekly visits with dressings also changed as needed. Patients were treated for a maximum of twelve weeks. Following twelve weeks of treatment, 18 of 37 patients treated with Oasis (49%) had complete wound closure compared to 10 of 36 patients treated with Regranex (28%).22

Salgado, et.al. conducted a prospective controlled study comparing Oasis® Wound Matrix and Aquacel® Ag in the treatment of mid-partial thickness burns.23 Five patients with burns were treated simultaneously with both products in different areas. Full thickness biopsies of the treated areas were taken at zero and seven days. Burns treated with Oasis had higher epithelial maturation index (6.2 ± 0.84) compared to burns treated with Aquacel (3.2 ± 3.28). Oasis treated burns produced a lower score according to Vancouver Scar Scale (3.6 ± 2.6) when compared to Aquacel treated burns 7.2 ± 2.5). The authors concluded that ECM matrices favour the wound healing process.23

Efficacy of CAMPs as a class of medical devices is well established in the management of hard-to-heal wounds. This retrospective, single centre, non-comparative post-market study will retrospectively collect and evaluate real-world performance data specifically for InnovaMatrix® AC.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 years or older at the time the data were reported.
* Subjects with hard-to-heal wound(s), defined as those that have failed to show improvement (which is defined as ≥50% reduction in wound area) over 4-weeks of standard wound care.
* Initial Wound area that is >0.5 cm2 and <10 cm2
* InnovaMatrix® AC applied to target wound(s) for a minimum of two consecutive weekly visits inside a 4-week period.
* Subjects were compliant with wound protection strategies through treatment period (offloading, compression, etc).
* The target wound(s) is not undergoing active management at the time of data entry.

Exclusion Criteria:

* Wound area showed ≥50% reduction in 4-weeks preceding initial InnovaMatrix® AC application.
* Cases where InnovaMatrix® AC was not applied at a minimum of two consecutive weekly visits inside a 4-week period.
* Subjects who were non-compliant with additional wound protection strategies (offloading, compression, etc)
* Subjects with severe comorbidities that significantly impact healing ability, or ability for subject to be compliant with wound protection strategies, such as: peripheral vascular disease (ABI <0.4, >1.3)1, severely uncontrolled diabetes (Hgb A1C >9.0%), neurodegenerative disorders, Charcot foot, high dose corticosteroid or other immunosuppressant, etc
* Wound area <0.5 cm2 or >10 cm2
* The target wound is still under active treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects seen at the study site between 1 May 2022 (the date of first product use according to the study site) to 27 March 2024 (the date of contract signature), who meet the inclusion and exclusion criteria. There will be no new patient visits associated with this retrospective study, therefore patient duration is not applicable.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Percent Area Reduction | 4 months
  Percent area reduction of target wound area at 4 weeks compared to baseline will be listed and tabulated over all eligible subjects, as calculated by wound length multiplied by wound width.

SECONDARY OUTCOMES:
Time to Complete Wound Closure | 4 months
  Time to wound closure as recorded in days and calculated as the difference from baseline and the date of the first event that wound closure is recorded for all eligible subjects. Wound closure will be defined as the first time point at which both of the following occur: 1) A value of 76-100% is recorded for % epithelisation tissue in the Wound Assessment form, and 2) The area of the wound (as calculated in Section 7.1) is 0 cm2.
Percent Granulation Tissue | 5 months
  Percent granulation tissue and its change from baseline will be tabulated as a shift table over all eligible subjects comparing baseline to week 4, week 12, and week 20.
Change in percent epithelialisation tissue | 4 months
  The change in percent epithelisation tissue at each interval will be summarised for percent granulation tissue for all eligible subjects. For subjects that have completed the study and have healed prior to the timepoint being summarised, the percent epithelialisation tissue will be imputed at a value of 76-100

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dr Michaelis, DO, Principal Investigator — Charleston Wound Care Centre
Locations (1):
- Charleston Wound Care Centre, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized data extract